CLINICAL TRIAL: NCT04581837
Title: Predictors and Outcomes of Occlusion of Jailed Side Branches Following Main Vessel Coronary Artery Stenting
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Adel Mekawy, principal investigator, Assiut University
Other Study IDs: 2DSTEBIFURCATION
Record Dates: First submitted 2020-09-09; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 2D-speckle tracking echocardiography — Two-dimensional speckle tracking echocardiography (2D-STE) allows for an angle-independent evaluation of myocardial strain, and provides comprehensive information on LV myocardial contractility. Thus, 2DSTE is superior in detecting subtle deteriorations of contractility. we will take 2D speckle tracking views for LV and RV strain (4ch, 2ch, 3ch, RV modified view).

SUMMARY:
Assessment of possible predictors of occlusion of jailed side branches following main vessel coronary artery stenting and detection of clinical, electrocardiographic and echocardiographic changes following occlusion of jailed side branches postprocedural and at 3 months follow-up.

DETAILED DESCRIPTION:
Coronary bifurcation lesion (CBL) involves coronary artery stenosis adjacent to and/or including the origin of a significant side branch (SB) 1. Treatment of bifurcation lesions constitute about 15% of coronary interventions and are consequently of major clinical interest 2. Even in the modern era of per-cutaneous coronary intervention(PCI) with stent implantation, treatment of bifurcations is hampered by a higher event rate and requires longer procedure time, more radiation exposure, and higher volumes of contrast material compared with non-bifurcation lesions 3 .

Occlusion of large side branches (SBs) may result in significant adverse clinical events 4. Occlusion of jailed sizable septal and right ventricular (RV) side branches (non-classic bifurcations) is often overlooked following left anterior descending (LAD) and right coronary artery (RCA) main vessel stenting, respectively. Most of the operators decline intervening in these side branches on contrary to classic bifurcations as diagonals and obtuse marginal branches, for example. Whether or not intervening with these occluded jailed side branches have clinical implications or even sub clinical left ventricular (LV) dysfunction was not previously elucidated and warrants studying.

Left ventricular function is an important predictor of outcome in patients with coronary artery disease (CAD). Extensive myocardial ischemia can cause decreased LV contractility and function 5. Conventional echocardiography enables us to identify significant left ventricular dysfunction but not sub-clinical dysfunction [10]. Two-dimensional speckle tracking echocardiography (2D-STE) allows for an angle-independent evaluation of myocardial strain, and provides comprehensive information on LV myocardial contractility. Thus, 2DSTE is superior in detecting subtle deterioration of contractility 6 .

In this study, investigators tried to explore the possible predictors and outcomes following occlusion of jailed side branches after main vessel coronary artery stenting, in both classic and non-classic bifurcations, and whether intervening via various techniques would have clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to cathlab for elective PCI along one year duration
* patients who have significant main vessel lesion subtending large, sizable (≥2mm) side branches (Medina 1,0,0 / 1,1,0 / 0,1,0)

Exclusion Criteria:

* acute myocardial infarction
* previous CABG
* LV EF<50%
* baseline SWMA in the territory of the vessel to be stented
* totally occluded main vessel.
* small (<2mm) side branch
* any ostial, mid or distal significant side branch disease at baseline.
* true bifurcation lesions (Medina 1,0,1 / 1,1,1 / 0,1,1) with upfront 2-stent strategy.
* advanced renal impairement

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting for elective PCI will undergo 2D-STE before the procedure and if found to have bifurcation lesion will undergo 2D-STE within 24 hours after the procedure and after 3 months
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Detection of changes in sub-clinical LV dysfunction after elective PCI to bifurcation lesions by detecting changes in LV global and regional longitudinal strain by 2D-speckle tracking echocardiography. | post-procedural (immediately after procedure) and at 3-months follow-up

SECONDARY OUTCOMES:
Detection of peri-procedural myocardial injury (PMI) | within 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Youssif, Doctorate, Study Director — Assiut University

REFERENCES:
- [Background] Yurtdas M, Asoglu R, Ozdemir M, Asoglu E. An Upfront Two-Stent Strategy for True Coronary Bifurcation Lesions with A Large Side Branch in Acute Coronary Syndrome: A Two-Year Follow-Up Study. Medicina (Kaunas). 2020 Feb 29;56(3):102. doi: 10.3390/medicina56030102. PMID 32121323
- [Background] Palinggi BP, Firman D. Carina Bifurcation Angle and Side Branch Occlusion in Coronary Bifurcation Lesions Intervention: Angiographic Lesions Characteristic Role in Determining Its Relation. Int J Angiol. 2019 Jun;28(2):137-141. doi: 10.1055/s-0038-1676042. Epub 2018 Nov 29. PMID 31384112
- [Background] Tsuchida K, Colombo A, Lefevre T, Oldroyd KG, Guetta V, Guagliumi G, von Scheidt W, Ruzyllo W, Hamm CW, Bressers M, Stoll HP, Wittebols K, Donohoe DJ, Serruys PW. The clinical outcome of percutaneous treatment of bifurcation lesions in multivessel coronary artery disease with the sirolimus-eluting stent: insights from the Arterial Revascularization Therapies Study part II (ARTS II). Eur Heart J. 2007 Feb;28(4):433-42. doi: 10.1093/eurheartj/ehl539. Epub 2007 Jan 31. PMID 17267457
- [Background] Zhang D, Xu B, Yin D, Li Y, He Y, You S, Qiao S, Wu Y, Yan H, Yang Y, Gao R, Dou K. Predictors and Periprocedural Myocardial Injury Rate of Small Side Branches Occlusion in Coronary Bifurcation Intervention. Medicine (Baltimore). 2015 Jun;94(25):e992. doi: 10.1097/MD.0000000000000992. PMID 26107685
- [Background] Mohamed Alsenbsey, Basem Asham, Sanaa Shaker Aly, Samar Sayed Ahmed, A. B. Role of insulin resistance in essential hypertensive patients in Qena Governorate, Egypt. Al-Azhar Assiut Med. J. 16, 99-104 (2018).
- [Background] Wang P, Liu Y, Ren L. Evaluation of left ventricular function after percutaneous recanalization of chronic coronary occlusions : The role of two-dimensional speckle tracking echocardiography. Herz. 2019 Apr;44(2):170-174. doi: 10.1007/s00059-017-4663-1. Epub 2018 Jan 16. PMID 29340717